CLINICAL TRIAL: NCT00265863
Title: Phase II Study of Laparoscopic Hyperthermic Peritoneal Chemotherapy for Malignant Ascites
Brief Title: Mitomycin as a Hyperthermic Peritoneal Perfusion in Treating Patients With Malignant Ascites
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Todd Tuttle, MD, Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS043
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Cancer
Keywords: malignant ascites
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Malignant Ascites (Experimental): Patients meeting protocol criteria enrolled with malignant ascites.
  Interventions: Drug: mitomycin C

INTERVENTIONS:
Drug: mitomycin C — Mitomycin C is infused into the abdominal cavity by hyperthermic perfusion over 60 minutes.
  Other Names: MTC

SUMMARY:
RATIONALE: Hyperthermia therapy kills tumor cells by heating them to several degrees above normal body temperature. Peritoneal infusion of heated chemotherapy drugs, such as mitomycin, may kill more tumor cells.

PURPOSE: This phase II trial is studying how well mitomycin works when given as a hyperthermic peritoneal perfusion in treating patients with malignant ascites.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of laparoscopic hyperthermic perfusion of mitomycin C in preventing relapse at 4 weeks post-treatment in patients with malignant ascites.

Secondary

* Determine any improvement in the quality of life of patients treated with this procedure.

OUTLINE: This is a nonrandomized study.

Patients undergo laparoscopic surgery to remove ascitic fluid and any intraabdominal adhesions and to place 2 inflow and 2 outflow catheters. Mitomycin C is infused into the abdominal cavity by hyperthermic perfusion over 60 minutes.

Quality of life is assessed at study entry and at 4 weeks.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peritoneal metastases and malignant ascites by physical examination, ultrasound, or CT scan
* Not eligible for cytoreductive surgery based on any of the following criteria:

  * Metastases outside peritoneal cavity
  * Poor performance status
  * Unresectable peritoneal disease
* Must have undergone at least 1 prior paracentesis procedure
* No ascites caused by any of the following conditions:

  * Cardiac failure
  * Nephrotic syndrome
  * Pancreatic ascites
  * Chylous ascites
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 70,000/mm^3
* Bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test

Exclusion Criteria:

* Prior peritoneal chemotherapy
* Dense intraabdominal adhesions limiting laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Prevention of malignant recurrence | Week 4 after treatment

SECONDARY OUTCOMES:
Quality of life after treatment | Week 4 after treatment
Comparison of serum vascular endothelial growth factor (VEGF) levels | Pretreatment and Week 4 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Tuttle, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States